CLINICAL TRIAL: NCT07112924
Title: CCM Technologies OPEN HF Registry: Observational Patient EvaluatioN of CCM® Therapy for Heart Failure
Brief Title: CCM OPEN HF Registry
Acronym: CCM OPEN HF
Status: Recruiting | Type: Observational
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Other Study IDs: OPEN_CA_CP_2025
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; CCM; Optimizer; Implantable Pulse Generator; FDA Approved; Heart Failure Hospitalization; Ischemic vs non-ischemic; CRT non-responders; Patients with concomitant devices; Patients with wide, intermediate, narrow QRS; Patients with cardiac amyloidosis
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Retrospective Cohort: Prospective Cohort
- Hybrid (Retrospective-Prospective) Cohort: Patients who will receive/ have received CCM therapy with an Impulse Dynamics devices
- Prospective Cohort: Patients who will receive CCM therapy with an Impulse Dynamics devices

SUMMARY:
The registry has been designed to evaluate the long-term safety and efficacy of CCM therapy in a real-world setting.

DETAILED DESCRIPTION:
This is a global, prospective and retrospective, multicenter, single-arm, observational study intended to include patients who will receive/have received CCM therapy with an Impulse Dynamics system, including future CCM technologies (e.g. CCM-D), for a follow-up period of at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have /will be implanted with Impulse Dynamics CCM technologies (e.g. CCM or CCM-D when available) as determined by investigators
* Willing and able to provide informed consent, including for use of data for research purposes (e.g. publication, sub-studies/sub-analyses)

Exclusion Criteria:

* Noncompliant patients (e.g. for follow-up visits, medication, etc.) as determined by investigators.
* Subjects with a mechanical tricuspid valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will receive/have received CCM therapy with an Impulse Dynamics system
Sampling Method: Probability Sample
Enrollment: 5500 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2035-08-15 (Estimated); Study Completion 2036-08-01 (Estimated)

PRIMARY OUTCOMES:
Assess CCM's effect on the rate and length of stay of heart failure (HF) hospitalizations | 1 Year
  Change in the HF hospitalization / urgent HF visit rate and hospital length of stay from 1 year prior to 1 year following index implantation.
Demonstrate the long-term safety of CCM therapy in a real-world setting, by assessing the rate of device- or procedure-related complications. | 5 Years
  Rate of freedom from a composite of device- or procedure-related complication post-index implantation procedure.
  Serious procedure related complications occurring through the end of 30 days following the index procedure.
  Serious CCM device-related complications* occurring through the end of 1-year following the index procedure.
  * excluding lead-related complications

SECONDARY OUTCOMES:
Assess CCM's effect on clinical outcomes | 5 Years
  Composite of all-cause mortality, heart-failure hospitalizations/urgent heart failure visits, progression to LVAD/heart transplant 1-, 3-, and 5-years following the index procedure.
Assess CCM's effect on mortality (all-cause, cardiovascular, and heart failure related) | 5 Year
  All-cause: Observed mortality will be compared to predicted mortality for the subject group according to the Seattle Heart Failure Model (SHFM) and/or Meta-analysis Global Group in Chronic Heart Failure (MAGGIC) at 1-, 3-, and 5-years following the index procedure.
  Cardiovascular related mortality will be assessed at 1-, 3-, and 5-years following the index procedure.
Assess CCM's effect on healthy days at home (HDAH) | 3 Years
  Assessment of HDAH 1 year prior to 3 years following index implantation.
Assess CCM's effect on functional capacity | 5 Year
  Change in NYHA Functional Class from baseline to 1-, 2-, 3-, 4-, and 5-years following the index procedure.
  Change in 6-minute walk test (6MWT) from baseline to 1 year following the index procedure.
Kansas City Cardiomyopathy Questionnaire (KCCQ) | 1 Year
  Change in KCCQ score from baseline to 6 months and 1 year after the index procedure. Scores range from 0 to 100, with higher scores showing better health status and lower scores showing worsen health status.
Assess CCM's effect cardiovascular reverse remodeling | 5 Year
  Change in LVEF, LVESV, LVEDV from baseline to 1-, 2-, 3-, 4-, and 5-years following the index procedure.
Assess CCM's effect QRS duration | 5 Years
  Change in QRS duration from baseline to 1-, 2-, 3-, 4-, and 5-years following the index procedure.
Assess CCM's systemic effects | 5 Years
  Change in eGFR and BNP from baseline to 1-, 2-, 3-, 4-, and 5-years following the index procedure.
Assess long-term CCM device-related adverse events and lead related events | 5 Years
  An assessment of the incidence of CCM device-related serious complications and non-serious CCM-device-related observations occurring during the 5-year period following the index procedure.
Assess the dose response of CCM therapy | 5 Year
  Correlation of CCM % and milliamp (mA) delivered with clinical outcomes and health status
Evaluate subject battery charging compliance | 5 Year
  Assess overall battery charging compliance defined as 60 minutes of charging per 10-day period between charging sessions (Expressed as percentage of compliant charging periods per subject over time e.g., number of compliant charging cycles ÷ total expected cycles × 100%).
Assess the effect of ancillary equipment on clinical outcomes | 5 Years
  Impact of ancillary equipment on clinical outcomes at 1- 2-, 3-, 4-, and 5-years following the index procedure. Including but not limited to:
  Lead type: style-driven lead, lumenless lead
  Guiding sheath/catheter
Assess CCM clinical outcomes by subject sub-groups | 5 Years
  Assess CCM effectiveness at various timepoints in sub-groups of interest, including but not limited to:
  Male vs female <65 vs ≥ 65-year-old Ischemic vs non-ischemic CRT non-responders Patients with concomitant devices (e.g. CRT, pacemaker, LBBP) Patients with wide, intermediate, narrow QRS Patients with cardiac amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Hong, Study Director — Impulse Dynamics; Lee Ming Boo, Study Director — Impulse Dynamics
Locations (1):
- Cardiovascular Associates of Mesa, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: No
The data are part of an ongoing commercial development program and are considered proprietary at this stage.

REFERENCES:
- See also: Sponsor of CCM Studies — https://impulse-dynamics.com